CLINICAL TRIAL: NCT05376033
Title: Outcome of Root Canal Treatments Obturated With Calcium Silicate Based Sealers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Fausto Zamparini, University of Bologna, University of Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUTENDOPROSP
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Endodontically Treated Teeth
Keywords: root canal treatment; healing rate; warm obturation technique; bioceramic sealer
MeSH Terms: conditions — Tooth, Nonvital | interventions — Root Canal Obturation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Premixed Sealer + Single cone (Experimental): Premixed flowable hydraulic calcium silicate sealer was applied with a a K File #15 that was inserted into the canal to reach the WL - 3mm and gently moved around the root canal walls. Then, gutta-percha points were gently inserted at the WL -0.5mm and compacted with lateral condensation/vertical condensation.
  Interventions: Other: root canal filling with Ceraseal sealer
- Premixed Sealer + Thermafil (Experimental): Premixed bioceramic sealer was applied and previously described. Pre-heated carrier was inserted in the canal at WL-0.5mm. The carrier excess was removed with a Thermacut bur.
  Interventions: Other: root canal filling with Ceraseal sealer
- Sealer + Thermafil (Other): Epoxy-resin-based sealer was mixed and immediately inserted into the root canal using a K File #15. Pre-heated carrier was inserted in the canal at WL -0.5mm. The carriers excess was removed with a bur.
  Interventions: Other: root canal filling with Ceraseal sealer

INTERVENTIONS:
Other: root canal filling with Ceraseal sealer — root canal filling with Ceraseal sealer

SUMMARY:
The clinical use of a flowable premixed calcium-silicate bioceramic sealer used in association with warm carrier-based/single-cone technique will be compared with epoxy resin-based sealer with carrier-based technique.

DETAILED DESCRIPTION:
Healthy consecutive patients (n= 109) requiring 141 root canal treatments were enrolled in this study and divided in 3 groups (Group 1: Ceraseal + single cone cold technique n=47. Group 2: Ceraseal + Carrier-based technique n=47. Group 3 AH Plus + Carrier based technique n=47).

Periapical X-rays were taken preoperatively, after root canal filling and after 6, 12 and 24 months. Two evaluators blindly assessed the Periapical Index (PAI) and sealer extrusion in the 3 groups (k =0.90). Healing rate and survival rate were also analysed.

Chi square tests was used to analyse significant differences among the groups. Multilevel analysis was performed to analyse the factors associated to healing status and survival status.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years
2. no use of antiresorptive or antiangiogenic drug
3. healthy status (ASA 1 or 2).
4. Needing one or more root canal treatment

Exclusion Criteria:

1. Teeth with less than 2 walls of structural integrity
2. Wide apexes (>40 diameter)
3. ASA > 3,
4. Any pathology that could compromise bone healing or the immune response,
5. pregnancy or breast feeding
6. heavy smoking (>15 cigarettes/day), (Tverdal & Bjartveit 2006)
7. exposure to radiation therapy focussed on the head and neck region and malignant disease directly involving the jaws.
8. Lacks of occlusal contacts

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Healing rate | 24 months
  Periapical index minor than 3 at the endline

SECONDARY OUTCOMES:
Survival rate | 24 months
  presence of root canal treated tooth at the endline

CONTACTS AND LOCATIONS:
Locations (1):
- Dental School University of Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No